CLINICAL TRIAL: NCT00229294
Title: Fibromyalgia in Men Suffering From PTSD
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA- 03-2925-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Fibromyalgia; Posttraumatic Stress Disorder; Major Depressive Disorder
MeSH Terms: conditions — Fibromyalgia; Stress Disorders, Post-Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Assessing FM and psychiatric state among PTSD, MDD and healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without any current or past psychiatric disorder
* Current diagnosis of PTSD
* Current diagnosis of MDD

Exclusion Criteria:

- Psychotic features

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2004-03; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University